CLINICAL TRIAL: NCT04831944
Title: A Phase 1, Open-Label Study to Evaluate the Pharmacokinetics and Safety of Parsaclisib in Participants With Normal Hepatic Function and Participants With Hepatic Impairment
Brief Title: To Evaluate the Safety, and Pharmacokinetics of Parscaclisib in Participants With Normal Hepatic Function and Hepatic Impairment.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INCB 50465-108
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Advanced Malignancies
Keywords: Hepatic Impairment; parsaclisib
MeSH Terms: interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Group 1 : Severe hepatic impairment (Experimental): Child Pugh (CP) assessment score of 10-14 points
  Interventions: Drug: parsaclisib
- Treatment Group 2 : Moderate hepatic impairment (Experimental): Child Pugh (CP) assessment score of 7-9 points
  Interventions: Drug: parsaclisib
- Treatment Group 3 : Mild hepatic impairment (Experimental): Child Pugh (CP) assessment score of 5-6 points
  Interventions: Drug: parsaclisib
- Treatment Group 4 : Normal hepatic impairment (Experimental): Normal hepatic function
  Interventions: Drug: parsaclisib

INTERVENTIONS:
Drug: parsaclisib — parsaclisib will be administered orally after 8 hours of fasting.
  Other Names: INCB050465

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics and safety of parsaclisib in participants With normal hepatic function and participants with hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with hepatic impairment.
* Participants eligible for Group 4 should be in good health.
* Participants eligible for Groups 1 through 3 may have medical findings consistent with their degree of hepatic dysfunction.
* Participants with abnormal findings considered not clinically significant by the investigator are eligible.
* Body mass index within the range of 18.0 to 40.0 kg/m2 (inclusive) at screening.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Evidence of rapidly deteriorating hepatic function.
* Participants with serum calcium and phosphorus levels over the upper limits of the institutional normal ranges.
* History or current diagnosis of uncontrolled or significant cardiac disease indicating significant risk of safety for participation in the study, including any of the following:
* Participants who have a current, functioning organ transplant or have a scheduled organ transplant in the next 6 weeks from check-in.
* History of malignancy within 5 years of screening, with the exception of cured basal cell carcinoma, squamous cell carcinoma of the skin, ductal carcinoma in situ, or Gleason 6 prostate cancer.
* History of clinically significant gastrointestinal disease or surgery (cholecystectomy and appendectomy are allowed) that could impact the absorption of study drug.
* Participants with severe ascites or an encephalopathy ≥ Grade 2.
* Any major surgery within 4 weeks of screening.
* Donation of blood to a blood bank within 4 weeks of screening (within 2 weeks for plasma only).
* Blood transfusion within 4 weeks of check-in. Current or recent history (within 30 days before screening) of a clinically significant bacterial, fungal, parasitic, or mycobacterial infection, or currently receiving systemic antibiotics. Current clinically significant viral infection at screening or check-in.
* Positive serology for hepatitis B virus (eg, hepatitis B surface antigen) or human immunodeficiency virus. Participants whose results are compatible with immunity due to infection or prior immunization for hepatitis B may be included at the discretion of the investigator.
* History of alcoholism within 3 months of screening.
* Positive breath test for ethanol or positive urine screen for drugs of abuse that is not otherwise explained by permitted concomitant medications.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) of study drug administration with another investigational medication or current enrollment in another investigational drug protocol.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) of study drug administration with strong or moderate inducer or potent inhibitor of CYP3A4.
* Receipt of live (including attenuated) vaccines or anticipation of need for such a vaccine during the study. (Note: Non-live or inactivated vaccines allowed up to 2 weeks before first dose administration.)
* Known hypersensitivity or severe reaction to parsaclisib or excipients of parsaclisib.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator. Inability to be venipunctured or tolerate venous access.
* Participants eligible for Group 4 who have a history or presence of liver disease or liver injury as indicated by an abnormal clinically significant liver function profile at screening or check-in.
* Participants eligible for Group 4 who have a positive test for hepatitis C virus.
* Participants eligible for Group 4 who used tobacco- or nicotine-containing products within 6 months of screening.
* Women who are pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Parameter : Cmax of parsaclisib | 5 Days
  Maximum Observed Plasma Concentration of parsaclisib
Pharmacokinetics Parameter : AUC 0-∞ of parsaclisib | 5 Days
  Area Under the Concentration-time Curve From 0 to Infinity of parsaclisib
Pharmacokinetics Parameter : AUC(0-t) of parsaclisib | 5 Days
  Area Under the concentration- time curve up to the last measurable concentration of parsaclisib

SECONDARY OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAE) | Up to10 Days
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Pharmacokinetics Parameter : tmax of parsaclisib | 5 Days
  Time to reach maximum plasma concentration of parsaclisib
Pharmacokinetics Parameter : t1/2 of parsaclisib | 5 Days
  Apparent terminal phase disposition half-life of parsaclisib
Pharmacokinetics Parameter : CL/F of parsaclisib | 5 Days
  Oral dose clearance of parsaclisib
Pharmacokinetics Parameter : Vz/F of parsaclisib | 5 Days
  Apparent oral dose volume of distribution of parsaclisib

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Inland Empire Liver Foundation, Rialto, California
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, Hialeah, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute Tli the Liver Institute of South Texas List Downtown Office, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency